CLINICAL TRIAL: NCT06513520
Title: Evaluation of Monocyte Expression of HLA-DR (mHLA-DR) in the Multi-pathological Elderly Subject in Geriatric Service
Brief Title: Evaluation of Monocyte Expression of HLA-DR (mHLA-DR) in Geriatric Service
Acronym: SENIOR HLA DR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0650; ID RCB (Other: 2024-A01573-44)
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Immune System
Keywords: Elderly patient; Immune system; mHLA DR; Immunosenescence; Multipathological subject
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A sample of blood (4mL EDTA tube and 4ml heparin tube)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients in acute medical situation: Patients over 75 with polypathology hospitalised in geriatric wards, in acute situation: for example, patients presenting with an infection, cardiac decompensation, a complicated fall, acute renal failure, any acute or decompensated cardiovascular pathology, any discovery of cancer that has not been stabilised.
  Interventions: Biological: Blood sampling
- Patients in stable medical situation: Patients over 75 with polypathology hospitalised in geriatric wards, in a stable situation: these are patients who have not had an episode of decompensation or infection for at least 7 days.
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Additional blood tube collection during routine blood sampling.

SUMMARY:
The acceleration of population aging and the improved management of comorbidities lead to an increase in the number of multi-pathological elderly patients admitted to geriatric services. This is an extremely specific population in terms of immunology due to the presence of immunosenescence (physiological aging of the immune system) and the potential additional effect of multiple chronic pathologies (comorbidities) presented by these patients.

The specific effect of multiple chronic pathologies on the immune status of elderly patients is currently underexplored because most studies on immune system aging only include elderly patients who do not have comorbidities or treatments that could impact the immune system (e.g. SENIEUR protocol). Therefore, their results are not applicable to patients in geriatric services.

The decrease in monocyte expression of HLA-DR (mHLA-DR) has been studied as a marker of immune alteration in intensive care units in the context of sepsis, but also in chronic pathologies (e.g. cancer, diabetes, renal insufficiency). These chronic pathologies are frequently found in elderly subjects.

The objective of the study would therefore be to investigate the relative contribution of age (immunosenescence) and comorbidities to the alteration of the immune status of geriatric patients through the measurement of mHLA-DR.

To date, no study has explored mHLA-DR in a population of multi-pathological geriatric patients. Our work aims to generate initial data through a pilot study in hospitalized multi-pathological subjects over 75 years old in geriatric services.

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* Patients aged over 75 hospitalised in one of the geriatric units defined as the research sites;
* Patient affiliated to a social security scheme;
* Patients or relatives who have been informed and have no objections to the research.

To be eligible in the acute situation sub-population:

- Patients presenting with an acute episode on admission or following a stay in the research sites; The acute episode is defined, for example, by an infection, cardiac decompensation, a complicated fall, acute renal failure, any acute or decompensated cardiovascular pathology, any discovery of cancer that has not been stabilised.

To be eligible in the stable situation sub-population:

- A patient who has not had an acute episode for at least 7 days.

Exclusion Criteria:

For all patients:

* Patients under legal protection: curatorship, guardianship, safeguard of justice ;
* Patients under exclusive comfort care for whom it has been decided not to take a blood sample;
* Patients undergoing long-term antibiotic treatment, i.e. with no defined stopping date;
* An immunocompromised patient or a patient undergoing immunosuppressive treatment (for example: HIV infection, a patient awaiting solid organ transplantation, a patient undergoing haematopoietic stem cell transplantation, a patient undergoing chemotherapy for a solid tumour or haematological malignancy, a patient suffering from an auto-immune disease and being treated with immunotherapy and/or immunosuppressive therapy and/or biotherapy, an asplenic or hyposplenic patient, a patient undergoing experimental potentially immunosuppressive treatment, a patient undergoing Eculizumab treatment, a patient presenting a hereditary immune deficiency).

For patients in an acute clinical situation:

- Patient previously included in the same sub-population.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study will focus on polypathological patients aged over 75 hospitalised in a geriatric ward.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
mHLA DR expression | up to 72 Hour
  Expression of mHLA DR assessed by flow cytometry and expressed as the number of antibodies bound per monocyte.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Dugoujon Hospital, Caluire-et-Cuire
  - Croix Rousse hospital, Lyon